CLINICAL TRIAL: NCT05963386
Title: An Open-Label, Non-Randomized, Single-Center, Investigator-initiated Phase II Trial to Determine the Efficacy and Safety of 177Lu-DOTA-EB-FAPI in Patients With Various End-stage Solid Tumors
Brief Title: Clinical Evaluation of 177Lu-DOTA-EB-FAPI in Patients With Various Solid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XMFHIIT-2023KY037
Record Dates: First submitted 2023-07-17; First posted 2023-07-27 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Refractory Solid Tumor
Keywords: Refractory solid tumor; Radioligand therapy; 177Lu-DOTA-EB-FAPI

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 177Lu-DOTA-EB-FAPI (Experimental): 177Lu-DOTA-EB-FAPI A maximum of 4 cycles of 90 mCi (3.3 GBq) 177Lu-DOTA-EB-FAPI, each. Route of administration: Slow intravenous infusion/injection (i.v.) Duration of treatment: 4 cycles, every 6 weeks
  Interventions: Drug: 177Lu-DOTA-EB-FAPI radionuclide therapy

INTERVENTIONS:
Drug: 177Lu-DOTA-EB-FAPI radionuclide therapy — radionuclide therapy using 177Lu-DOTA-EB-FAPI 90 mCi (3.3 GBq) will be performed 6-weekly. A maximum of 4 cycles will be administered.

SUMMARY:
Increased fibroblast activation protein expression is positively correlated with the aggressiveness of cancer. Radiolabeled fibroblast activation protein inhibitor therapy, also known as radioligand therapy has become a novel treatment for patients with refractory cancer and disease progression after multiple-lines treatment. However, a major problem in the therapeutic use of 177Lu-DOTA-FAPI has been its short half-life and fast rate of clearance. This study was designed to investigate the efficacy and safety of 177Lu-DOTA-EB-FAPI in patients with various solid tumors who had failed standard therapies.

DETAILED DESCRIPTION:
This investigator-initiated phase II study will include a maximum of 30 subjects with progressive cancer after multiple-line treatment, with an increased radiotracer uptake in tumors on 68Ga-FAPI-46 PET/CT. The fixed dose of 177Lu-DOTA-EB-FAPI is 3.3GBq (90 mCi) per cycle. Treatment is planned for up to 4 cycles, and the time interval between cycles is 6 weeks. The primary endpoint assessed the radiological response (according to RECIST criteria) after completion of radioligand therapy. The secondary endpoints included progression-free survival (PFS), overall survival (OS), dosimetry, and safety of 177Lu-DOTA-EB-FAPI.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and willingness to sign a written informed consent document.
* Age 18 and older.
* Confirmed unresectable or metastatic refractory cancer with measurable disease per RECIST (version 1.1) (i.e. at least 1 lesion > 1 cm or lymph node > 1.5 cm in short axis).
* Progressive disease after multiple-lines treatment.
* Completion of entry into 68Ga-FAPI-46 study and completion of scan. The tumor lesions showing increased radiotracer uptake on 68Ga-FAPI-46 PET/CT (defined as a maximum standardized uptake value ≥10 in more than 50% of metastatic lesions).
* Able to remain motionless for up to 30-60 minutes per scan.

Exclusion Criteria:

* Serum creatinine level >150 μmol/L.
* Hemoglobin level <8.0 g/dL; white-cell count < 2.0×109/L; platelet count < 50×109/L; total bilirubin level >3 times the upper limit of the normal range and serum albumin level <2.0 g/dL.
* Participants with Class 3 or 4 NYHA Congestive Heart Failure.
* Participants with severe allergy, or hypersensitivity to radiographic contrast material.
* Participants with claustrophobia.
* Pregnant or lactating women.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2024-09-15 (Actual); Study Completion 2024-10-05 (Actual)

PRIMARY OUTCOMES:
Radiological response (according to RECIST criteria) | 6 weeks, 12 weeks, 18 weeks, or up to 6 months
  RECIST objective response after completion of radioligand therapy, which was defined by response category between baseline and restaging after RLT. Disease control after RLT was defined as either complete response (CR), partial response (PR), or stable disease (SD). Disease control rate (DCR) was reported as the proportion of patients with disease control after RLT.

SECONDARY OUTCOMES:
Progression-free survival (PFS) and overall survival (OS) | disease progression, death or last follow-up conducted for all patients at the end of August 2024.
  PFS was recorded from start of RLT until RECIST progression, death, or last follow-up. OS was recorded from start of RLT until death or last follow-up conducted for all patients at the end of August 2024.
Dosimetry | 6 weeks
  Dosimetry, measured as the absorbed dose in tumors (Gy/GBq), was estimated in the first treatment cycle for each patient.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No